CLINICAL TRIAL: NCT00005726
Title: Evaluation of Low Literacy CVD Nutrition Education
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4935; R01HL046781 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To develop and evaluate a nutrition education program to reduce cardiovascular disease risk in persons with low literacy skills.

DETAILED DESCRIPTION:
BACKGROUND:

The setting for the study was the Minnesota Extension Service's Expanded Food and Nutrition Education Program (EFNEP), which was a U.S. Department of Agriculture-funded program to improve the nutrition knowledge and behavior of low-income individuals who were responsible for food preparation. The emphasis of EFNEP was on obtaining adequate and nutritious foods, and not on dietary behaviors for the prevention of chronic disease. Because a large proportion of this population had no more than an 8th grade education (30.9 percent nationally), EFNEP provided access to individuals with low literacy skills and a need for nutrition education for disease prevention. For example, a pilot study indicated that 34 of 42 respondents had never had their blood cholesterol level checked.

The study was part of an NHLBI initiative on "CVD Nutrition Education for Low Literacy Skills". The initiative originated within the Prevention and Demonstration Branch of the DECA, was approved by the September 1988 National Heart, Lung, and Blood Advisory Council, and released in July 1990.

DESIGN NARRATIVE:

The study developed education strategies using focus groups of both the Minnesota Extension Service's Expanded Food and Nutrition Education Program (EFNEP) program participants and the EFNEP paraprofessionals who delivered the program. The intent of the focus groups was to identify concerns, interests, barriers, and perceived needs for nutrition education for cardiovascular disease prevention. This information was used to develop effective education strategies that addressed the needs of the study participants, while accomplishing the study goal of effecting dietary change (specifically, decrease in dietary fat and cholesterol intake) for cardiovascular disease risk reduction.

The effectiveness of the nutrition education program was evaluated in a randomized trial, with pre- and post-intervention measures of dietary fat intake and plasma total and HDL cholesterol as outcome measures. The study was conducted in Hennepin, Ramsey and Dakota Counties, which had a total adult EFNEP enrollment of about 1,842 people. Because EFNEP enrollment was predominantly female (94 percent), this study was limited to adult women, age 18 or older. All 22 EFNEP paraprofessionals in these counties were randomized to intervention and control group. Randomization was at the level of paraprofessional to simplify program delivery and to minimize contamination between intervention and control groups. The differential changes in fat intake and plasma cholesterol level between the intervention and control groups were estimated using analysis of covariance, adjusting for within paraprofessional correlation and other potential confounders.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 1995-05 (Actual)

REFERENCES:
- [Background] Hartman TJ, McCarthy PR, Park RJ, Schuster E, Kushi LH. Results of a community-based low-literacy nutrition education program. J Community Health. 1997 Oct;22(5):325-41. doi: 10.1023/a:1025123519974. PMID 9353681
- [Background] Hartman TJ, McCarthy PR, Park RJ, Schuster E, Kushi LH. Focus group responses of potential participants in a nutrition education program for individuals with limited literacy skills. J Am Diet Assoc. 1994 Jul;94(7):744-8. doi: 10.1016/0002-8223(94)91940-2. PMID 8021415